CLINICAL TRIAL: NCT02530918
Title: Phase I Dose Escalation and Expansion Study of DS-7080a in Subjects With Neovascular Age-related Macular Degeneration or Diabetic Macular Edema
Brief Title: Study of DS-7080a for the Treatment of Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS7080-A-U101
Record Dates: First submitted 2015-08-17; First posted 2015-08-21 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Neovascular Age-Related Macular Degeneration; Diabetic Macular Edema
Keywords: DS-7080a Monoclonal Antibody
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Intervention Model Description: Sequential Assignment with 3 cohorts in Part 1, Parallel Assignment with 3 arms in Part 2, and Parallel Assignment with 2 arms in Part 3
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1 DS-7080a dose escalation (Experimental): 3 sequential ascending dose levels (1.0, 2.0, 4.0 mg), every 4 weeks for 12 weeks
  Interventions: Drug: DS-7080a
- Part 2 DS-7080a (Experimental): Specific dose (either the maximum tolerated dose or 4.0 mg) of DS-7080a determined in Part 1, every 4 weeks for 12 weeks
  Interventions: Drug: DS-7080a
- Part 2 ranibizumab (Active Comparator): Ranibizumab 0.5 mg, every 4 weeks for 12 weeks
  Interventions: Drug: Ranibizumab
- Part 2 DS-7080a and ranibizumab (Experimental): Specific dose of DS-7080a determined in Part 1 and ranibizumab 0.5 mg, every 4 weeks for 12 weeks
  Interventions: Drug: DS-7080a; Drug: Ranibizumab
- Part 3 DS-7080a (Experimental): Specific dose of DS-7080a determined in Part 1, every 4 weeks for 12 weeks
  Interventions: Drug: DS-7080a
- Part 3 ranibizumab (Experimental): Ranibizumab 0.3 mg, every 4 weeks for 12 weeks
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: DS-7080a — 1.0, 2.0, or 4.0 mg administered by a 50 μL intravitreal (IVT) injection of solution
  Other Names: Investigational product
  Arms: Part 1 DS-7080a dose escalation; Part 2 DS-7080a; Part 2 DS-7080a and ranibizumab; Part 3 DS-7080a
Drug: Ranibizumab — 0.3 mg or 0.5 mg administered by a 50 μL IVT injection of solution
  Other Names: Lucentis
  Arms: Part 2 DS-7080a and ranibizumab; Part 2 ranibizumab; Part 3 ranibizumab

SUMMARY:
The purpose of this study is to test DS-7080a, a monoclonal antibody, as a new treatment for neovascular age-related macular degeneration (AMD) and diabetic macular edema (DME). The hypothesis of the study is that DS-7080a is safe and shows preliminary efficacy in patients with these conditions either alone or in combination with ranibizumab. This study is organized into 3 Parts: Part 1 Dose Escalation in AMD participants, Part 2 Dose Expansion in AMD participants, and Part 3 Dose Expansion in DME participants.

In Part 1, participants will be enrolled into 3 sequential, ascending dose-level cohorts in non-randomized uncontrolled manner with the main purpose to determine the recommended dose.

In Part 2, participants will be randomized to 1 of 3 arms of either monotherapy with DS-7080a or monotherapy with ranibizumab, which is an active control, or combination therapy of DS-7080a plus ranibizumab (ranibizumab will be administered 30 minutes prior to DS-7080a).

In Part 3, subjects with DME will be assigned to 1 of 2 arms of either monotherapy with DS-7080a or monotherapy with ranibizumab. DS-7080a or ranibizumab will be administered 3 times: on Baseline/Day 1, Day 29, and Day 57.

Both Parts 2 and 3 will consist of 8 visits including a 14-day screening phase, an 84-day treatment period, and a 28-day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

For parts 1 and 2:

* ≥ 50 years of age
* Has active primary subfoveal choroid neovascularization (CNV) lesions secondary to age-related macular degeneration (AMD)
* CNV ≥ 50% of total lesion size in study eye
* Central sub-field thickness > 315 µm on spectral domain optical coherence tomography (SD-OCT) in the study eye
* Has BCVA letter score required at screening visit:
* For Part 1, ≤ 49 (approximately 20/100 or worse) in the study eye and ≥ 49 (approximately 20/100 or better) in the fellow eye
* For Part 2, 78 to 25 (approximately 20/32 to 20/320) in the study eye

For Part 3:

* Is ≥ 18 years of age with retinal thickening due to diabetic macular edema (DME)
* Has central sub-field thickness (CST) > 335 μm in the study eye
* Has BCVA letter score at screening visit 78 to 25 letters (approximately 20/32 to 20/320) in the study eye

Exclusion Criteria:

For Parts 1 and 2:

* Has used any long acting steroids, either systemically or intraocularly, within 6 months of Baseline Visit
* Has total lesion size > 12 disc areas (30.5 mm2) in the study eye
* Has presence of retinal pigment epithelial tears or rips involving the macula in the study eye
* Has history of any vitreous hemorrhage within 4 weeks prior to Screening Visit in the study eye
* Has presence of causes of CNV other than AMD
* Had prior vitrectomy in the study eye
* Has history of retinal detachment or treatment or surgery for retinal detachment in the study eye
* Has any history of a full thickness macular hole in the study eye
* Had any intraocular or periocular surgery within 3 months of Baseline Visit on the study eye, except lid surgery
* Has uncontrolled glaucoma in the study eye
* Has active intraocular inflammation or periocular infection in either eye
* Has any history of uveitis in either eye of scleromalacia in either eye
* Has aphakia or pseudophakia in the study eye
* Had previous therapeutic radiation in the region of the study eye
* Has history of corneal transplant or corneal dystrophy in the study eye
* Has significant media opacities in the study eye (e.g. cataract) that could require either medical or surgical intervention during the study period
* Is a women who is pregnant, breastfeeding, or of childbearing potential and unwilling to practice two measures of adequate contraception throughout the study

For Part 1 only:

* Had any ocular (in the study eye) or systemic treatment or surgery for neovascular AMD within 4 weeks of Baseline Visit, except dietary supplements or vitamins
* Has a subretinal hemorrhage that is ≥ 50% of the total lesion area in the study eye
* Has scarring or fibrosis, making up >50% of total lesion or involving the center of the fovea in the study eye

For Part 2 only:

* Had any prior therapy in the study eye within 3 months of Baseline Visit, except dietary supplements or vitamins

For Part 3:

* Has used any steroids, either systemically or ocular in the study eye (other than fluocinolone), within 6 months of Baseline Visit
* Has macular edema in the study eye considered to be due to a cause other than DME
* Has high-risk proliferative diabetic retinopathy (PDR) in the study eye
* Has decrease in BCVA in the study eye due to causes other than DME
* Has significant macular ischemia in the study
* Has choroidal neovascularization (CNV) secondary to any etiology
* Has retinal pigment epithelial tears or rips involving the macula in the study eye
* Had any vitreous hemorrhage within 4 weeks prior to Screening/Visit 1 in the study eye
* Had prior vitrectomy in the study eye
* Has history of retinal detachment or treatment or surgery for retinal detachment in the study eye
* Has history of a full thickness macular hole in the study eye
* Had any intraocular or periocular surgery within 3 months of Baseline Visit
* Has uncontrolled glaucoma in the study eye
* Had prior trabeculectomy or other filtration surgery in the study eye
* Has active intraocular inflammation or periocular infection in either eye
* Has current or history of scleromalacia in either eye
* Has aphakia or pseudophakia with absence of posterior capsule
* Has previous therapeutic radiation in the region of the study eye
* Has history of corneal transplant or corneal dystrophy in the study eye
* Has concurrent ocular condition in the study eye which, in the opinion of the investigator, could either increase the risk to the subject beyond what is to be expected from standard procedures of intraocular injection, or which otherwise may interfere with the injection procedure or with evaluation of safety, tolerability, or efficacy
* Has systolic blood pressure ≥160 mmHg and/or a diastolic blood pressure ≥95 mmHg at Screening
* Has an estimated Glomerular Filtration Rate (eGFR) of < 15 mL/min/1.73 m^2 as per the creatinine equation (CKD-EPI) at Screening
* Has any history of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications
* Is a women who is pregnant, breastfeeding, or of childbearing potential and unwilling to practice two measures of adequate contraception throughout the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing any treatment-emergent adverse event (TEAE) | 16 weeks
  Treatment-emergent AEs (TEAEs) are defined as those adverse events (AEs) that were new or got worse between the start of study treatment and the end of the follow-up period.
Best Corrected Visual Acuity (BCVA) score | 12 weeks
  Visual acuity of both eyes will be assessed at all study visits using the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score. The patient starts are the top of the chart and begins to read down the chart. The patient reads down the chart until he or she reaches a row where a minimum of three letters on a line cannot be read. The patient is scored by how many letters could be correctly identified. Added to the score for the last row where the participant could read all five letters correctly are scores for each additional letter that could be read correctly in the next row. This is the BCVA score. A higher score means better visual acuity (sharpness of vision).

SECONDARY OUTCOMES:
Change from baseline in retinal thickness and volume | 12 weeks
  Retinal thickness and volume are assessed by spectral domain optical coherence tomography (SD-OCT)
Change from baseline in retinal leakage | 12 weeks
  Retinal leakage is assessed by fluorescein angiography (FA)
Plasma concentrations | 12 weeks
  Concentration of study drug in blood plasma
Part 3 only: Change from baseline in vessel flow density, foveal avascular zone (FAZ) area, and FAZ shape | 12 weeks
  Vessel flow density, foveal avascular zone (FAZ) area, and FAZ shape are assessed by OCT angiography (OCT-A)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (12):
- United States (12):
  - Phoenix, Arizona
  - Arcadia, California
  - Beverly Hills, California
  - Palm Desert, California
  - Fort Myers, Florida
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Omaha, Nebraska
  - Abilene, Texas
  - Austin, Texas
  - San Antonio, Texas
  - Silverdale, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at http://www.clinicalstudydatarequest.com. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://www.clinicalstudydatarequest.com/Study-Sponsors-DS-Details.aspx
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received EU and US marketing approval on or after 01 January 2014 or by the US or EU Health Authorities when regulatory submissions in both regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States and the European Union from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://www.clinicalstudydatarequest.com/Study-Sponsors-DS-Details.aspx